CLINICAL TRIAL: NCT02172989
Title: Clinical Application of Near-infrared Fluorescence Guided Localization on Breast Surgery in Benign Breast Neoplasm ; Observational Pilot Study for 20 Patients.
Brief Title: Clinical Application of Near-infrared Fluorescence Guided Localization on Breast Surgery in Benign Breast Neoplasm.
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, So-Youn Jung, Medical Dotor, National Cancer Center, Korea
Other Study IDs: NCC-1410202-1
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Benign Breast Neoplasm
Keywords: Near-infrared fluorescence; Indocyanine green, ICG; Radio-guided surgery; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Near-infrared (NIR) fluorescence imaging using indocyanine green (ICG) has been used for breast cancer surgery such as sentinel lymph node (SLN) mapping and breast cancer localization.

In this study, our hypothesis are as following:

1. As inject only indocyanine green (ICG), it provide the surgeon visual guidance to ensure better outcome.
2. indocyanine green (ICG) permitted accurate preoperative and intraoperative detection of the SLNs as well as nonpalpable benign brest lesion in patients with breast cancer.

DETAILED DESCRIPTION:
Indocyanine green, ICG (ICG-fluorescence)

* ICG is the most commonly used fluorophore which approve by FDA.
* NIR-F imaging with ICG could be used in various surgeries. For example, SLN mapping in breast cancer and localization of liver metastasis, especially superficial lesion
* Contains sodium iodide, patients who have history of allergy to iodides should be used as caution.

Nonpalpable benign brest lesion localization

* New method for the localization and resection of non-palpable breast lesions.
* The breast lesion was correctly localized, and the area of ICG corresponded well to the site of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* nonpalpable benign breast lesion ≤ 2cm in patients with breast cancer.
* patients who need breast biopsy as treatment for breast cancer.
* Eastern Cooperative Oncology Group Performance status 0 or 1
* consented patients with more than 20 years, less than 70 years

Exclusion Criteria:

* nonpalpable benign breast lesion ≥ 2cm in patients with breast cancer.
* pregnancy
* history of severe allergy to ICG(Indocyanine Green)
* iode hypersensitiveness

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nonpalpable benign breast lesion ≤ 2cm in patients with breast cancer.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
non-palpable lesion localization rate | up to 6month
  non-palpable lesion localization rate = number of patients complete excision of lesion / 20 enrolled patients

SECONDARY OUTCOMES:
lesion of resection size, completeness of resection | up to 6month
  actual lesion of width*height*length / resection lesion of width*height*length

OTHER OUTCOMES:
physical assess | following up a week to 6 month
  number of patients with pigmented skin lesion, number of patients with complication, number of patients with breast lymphedema, number of patients with residual breast lesion using breast ultrsound

CONTACTS AND LOCATIONS:
Overall Officials: So-Youn Jung, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea